CLINICAL TRIAL: NCT01993576
Title: Histological Study of the (Intravenously Injected) ICG Distribution in Tumor Bearing Breasts and in Axillary Pieces of Dissection.
Brief Title: ICG Distribution Using NIF Imaging After IV Injection of ICG in Benign and Malignant Breast Cancer Tissue.
Acronym: EC2075
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-000100-41
Record Dates: First submitted 2013-05-06; First posted 2013-11-25 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer.
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- indocyanine green (Experimental): Indocyanine green is injected intravenously.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Intravenous injection of 0.25 mg/kg Indocyanine Green (ICG) before the surgery
  Other Names: ICG

SUMMARY:
The purpose of this study is to determine if NIF fluoresent imaging is an effctive approch to detect the margine of the breast tumoral tissue.

DETAILED DESCRIPTION:
Primary objective:

Definition of the histological distribution (intravascular, extra vascular, in specific cells) of ICG (pre-operatively intra-venously injected) at the level of tumoral and healthy tissues of breast cancer patients (and the potential of axillary lymph nodes found fluorescent).

Secondary objectives:

Evaluation of the ability of the fluorescence imaging to determine the tumor volume and, more specifically, the boundaries of tumor tissues which will be analyzed by the pathologist.

Analysis of the correlation between fluorescence and "margins" as defined operatively as tumor (microscopically by the pathologist).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological diagnosis of breast cancer for which a mastectomy with axillary dissection is planned.
* Informed Consent signed.

Exclusion Criteria:

* Diagnosis of breast cancer established by lumpectomy or "macro-biopsy".
* Operation after neo-adjuvant chemotherapy,
* Age less than 18 years.
* For pre-menopausal women, an operation planned for the second phase of their cycle.
* Inability to give informed consent.
* History of allergy or hypersensitivity to the investigational product, iodine.
* Clinical or biological hyperthyroidism.
* Known "toxic" thyroid nodules or known autonomous (hyperfunctional) thyroid.
* A reported pathological coronary artery disease.
* Creatinine > 1.5 mg / dl.
* During the 2 weeks before surgery, being on medications which are known to interfere with the ICG (ie anticonvulsants, heparin and haloperidol).
* Pregnancy or breast feeding period.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Study of the evantual difference of indocyanine in mammalian tissue in patients mastocmemezied for breast canrcinoma. | 10 months
  Detecting of the fluorescence in between benign and malignant tissue by near infra-red imaging with a camera dictated to identify the margin of the tumor, and Histological detection of indocyanine green distribution in tumor bearing breasts and in axillary pieces of dissection and the detection of tumor cells in lymphe nodes.

SECONDARY OUTCOMES:
Microscopical detection of indocyanine green in breast tissue. | 10 months.
  Detecting the fluorescence in between benign and malignant tissue by a microscope with a filter for near ifra-red at a good wave length of ICG.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Nogaret, Prof., Study Chair — Jules Bordet Institute; Isabelle Veys, MD, Study Chair — Jules Bordet Institute; Sophie VanKerckhove, biologist, Study Chair — Jules Bordet Institute; Philippe De Neubourg, MD, Study Chair — Jules Bordet Institute; Danielle Noterman, MD, Study Chair — Jules Bordet Institute
Locations (1):
- Jules Bordet Insitute, Brussels, Belgium, Belgium